CLINICAL TRIAL: NCT04383236
Title: Evaluation of the Effect of Probiotic Lozenges in the Treatment of Recurrent Aphthous Stomatitis: a Randomized, Controlled Clinical Trial
Brief Title: Probiotic Lozenges for Treatment of Recurrent Aphthous Stomatitis
Acronym: RAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reham Lotfy Aggour (Other)
Responsible Party: Sponsor-Investigator, Reham Lotfy Aggour, Associate professor of Oral Medicine, diagnosis & Periodontology, October 6 University
Organization: October 6 University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-2016
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Oral Ulcer
Keywords: Aphthous, lactobacillus, probiotics
MeSH Terms: conditions — Oral Ulcer | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: The study is a randomized, controlled, clinical trial
Who Masked: Outcomes Assessor
Masking Description: All clinical outcome variables are recorded by a single investigator whom is blinded to the treatment modalities
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ChocBalls (Experimental): (L. acidophilus containing lozenges, PharmaCare Europe Ltd; West Sussex, RH10 9NQ, UK)
  Interventions: Other: Probiotics
- Oracure oral gel (15 gm, Amun pharmaceutical company, Egypt) (Active Comparator): Each 100 g contains:
  Lidocaine HCI 2.0g. Cetylpyridinium chloride 0.1 g.
  Interventions: Drug: Oracure oral gel

INTERVENTIONS:
Other: Probiotics — Sixty adult (group A) and 60 children patients (group B) with diagnosis of minor RAS were included. Both groups were divided into two subgroups, AI and BI (test subgroups) and AII and BII (control subgroups). For test subgroups, probiotic lozenges were consecutively administered twice daily, for five days. The size and pain level of ulcers were recorded on treatment days 0, 3 and 5. The outbreak frequency of RAS within 6 months was investigated for all subgroups.
  Arms: ChocBalls
Drug: Oracure oral gel — Sixty adult (group A) and 60 children patients (group B) with diagnosis of minor RAS were included. Both groups were divided into two subgroups, AI and BI (test subgroups) and AII and BII (control subgroups). For control subgroups, oracure gel were consecutively applied twice daily, for five days. The size and pain level of ulcers were recorded on treatment days 0, 3 and 5. The outbreak frequency of RAS within 6 months was investigated for all subgroups.
  Arms: Oracure oral gel (15 gm, Amun pharmaceutical company, Egypt)

SUMMARY:
The application of host-modulating bacteria for therapeutic purposes is one of the strongest emerging fields. Probiotics are live microorganisms, which, when administered in an adequate amount, confer a health benefit on the host The study aimed to explore the effectiveness of probiotics in the treatment of the common ulcerative condition; minor recurrent aphthous stomatitis (RAS). We included sixty adult (group A) and 60 children patients (group B) with diagnosis of minor RAS . Both groups were divided into two subgroups, AI and BI (test subgroups ) and AII and BII (control subgroups). For test subgroups, probiotic lozenges were consecutively administered twice daily, for five days. The size and pain level of ulcers were recorded on treatment days 0, 3 and 5. The outbreak frequency of RAS within 6 months was investigated for all subgroups.

DETAILED DESCRIPTION:
The study aimed to explore the effectiveness of probiotics in the treatment of minor recurrent aphthous stomatitis (RAS). We performed a randomized, controlled clinical study. Sixty adult (group A) and 60 children patients (group B) with diagnosis of minor RAS were included. Both groups were divided into two subgroups, AI and BI (test subgroups) and AII and BII (control subgroups). For test subgroups, probiotic lozenges were consecutively administered twice daily, for five days. The size and pain level of ulcers were recorded on treatment days 0, 3 and 5. The outbreak frequency of RAS within 6 months was investigated for all subgroups. Compared to baseline, an improvement was evident for all subgroups. However, for effectiveness in pain reduction, a statistically significant difference in favor of AI was observed for all evaluation periods when compared to control subgroup. Regarding effectiveness in ulcer size reduction, a statistically significant difference in favor of BI was observed at day 5 when compared to control subgroup. No significant difference was observed in the effectiveness index between subgroups AI and BI (test subgroups) except in effectiveness in pain reduction at day 3. The outbreak frequency decreased significantly in subgroup BI. We concluded that topical application of probiotics decreased pain intensity and accelerate RAS healing. The effectiveness in pain reduction is more evident in adult patients while acceleration of healing is more evident in children. Probiotics could be a well-tolerated, topical therapeutic agent in the treatment of minor RAS

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18-45 years old, 2. Patients presenting with RAS with the following characteristics: a. Minor aphthous ulcers less than 48 hours' duration prior to enrolment, b. Size no greater than 10 mm in diameter, c. A history that ulcers normally more than 5 days to resolve without treatment. The inclusion criteria for group B is the same except age, children with RAS aged between 3 and 12 years were recruited for the study.

Exclusion Criteria:

* A known history of hypersensitivities, immunologic or systemic diseases, pregnancy, smoking,
* treatment with systemic steroid or other immunomodulatory agents within 1 month before the study
* use of nonsteroidal anti-inflammatory drugs or oral antihistamines within 1 month prior to the study
* treatment of the ulcer with any preparation or medication within 72 hours prior to the study
* treatment with systemic antibiotics within 2 weeks prior to the study and a history of adverse reactions to lactose or fermented milk products.
* Children with a positive family history of RAS were excluded.

Ages: 3 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-10-20 (Actual); Study Completion 2019-04-21 (Actual)

PRIMARY OUTCOMES:
Ulcer size reduction | 5 days
  The index ulcer's size was measured on treatment days 0, 3 and 5. The investigators measured the maximum and minimum diameters when the ulcer has an oval shape, using a calibrated dental probe with millimeter markings. The two measurements were then be multiplied to represent the cross-sectional areas of the ulcer.
Ulcer pain moderation | 5 days
  a visual analog scale (VAS) consisting of a 10-cm horizontal line between poles connoting no pain (origin) to unbearable pain was used. Subjects was told to mark the line with a vertical line at the point that best represented the present pain level of the ulcer

SECONDARY OUTCOMES:
Outbreak frequency/ 6 months | 6 months
  Participants were asked to estimate the average duration of episodes during the past 6 months and the potential to reduce the outbreak frequency of RAS within the next 6 months was investigated

CONTACTS AND LOCATIONS:
Overall Officials: Reham Aggour, Dr, Principal Investigator — Oral Medicine & Periodontology department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamal Y, Abdelwhab A, Salem ST, Fakhr M. Evaluation of the efficacy of supplementary probiotic capsules with topical clobetasol propionate 0.05% versus topical clobetasol propionate 0.05% in the treatment of oral lichen planus (a randomized clinical trial). BMC Oral Health. 2025 Mar 5;25(1):344. doi: 10.1186/s12903-024-05246-x. PMID 40045332
- [Derived] Aggour RL, Mahmoud SH, Abdelwhab A. Evaluation of the effect of probiotic lozenges in the treatment of recurrent aphthous stomatitis: a randomized, controlled clinical trial. Clin Oral Investig. 2021 Apr;25(4):2151-2158. doi: 10.1007/s00784-020-03527-7. Epub 2020 Aug 20. PMID 32820431

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT04383236/Prot_SAP_000.pdf